CLINICAL TRIAL: NCT03042559
Title: The Effects of Protonics Knee Brace Versus Hamstring Resisted Exercise on Individuals With Patellofemoral Pain Syndrome
Brief Title: Protonics Knee Brace Versus Hamstring Resisted Exercise (HRE) on Individuals With Patellofemoral Pain Syndrome
Acronym: HRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Everett Lohman, Professor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5160417
Record Dates: First submitted 2017-01-30; First posted 2017-02-03 (Estimated); Results first posted 2019-11-22 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-04

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Protonics knee brace (Active Comparator): All subjects were fitted with a regular-sized Protonics knee brace with resistive settings to resist knee flexion.
  Interventions: Device: Protonics Knee brace
- Sport cords (Experimental): Resistive sports cord to resist knee flexion.
  Interventions: Device: Sports Cords

INTERVENTIONS:
Device: Protonics Knee brace — The Protonics system has been introduced to physical therapists as a potential treatment for PFPS. The system includes a brace set to resist knee flexion and a set of specific exercises to perform daily. Through resistance to knee flexion, the system is advertised to decrease retropatellar contact pressure due to changes in pelvis inclination and available hip rotation. Specifically, resistance to knee flexion is purported to increase hamstring activity and inhibit the activity of the tensor fasciae latae and psoas muscles. The manufacturer asserts that prolonged use of the system results in greater hamstring activation, which leads to permanent structural changes through reciprocal inhibition at the hip and pelvis. The warm-up consisted of the subject wearing the ProtonicsTM knee brace set at a moderate resistance level and flexing the knees while sitting, standing, and reclining in the supine and prone positions.
  Arms: Protonics knee brace
Device: Sports Cords — Subjects assigned to the sport cord group were asked to do the same warm-ups and exercises using the sport cord in the supine, standing, sitting, and prone positions. prone. The only difference is that subjects were asked to only walk backwards instead of forwards in order to avoid activation of the hip flexor muscle. The appropriate level of resistance for each subject was calculated by multiplying their weight in pounds by 0.3. Subjects were then given either light, medium, or heavy resistance cords according to the following classification scheme: light (pink color) with resistance 3 (R3), 0-30 lbs.; medium (orange color) with resistance 5 (R5) 0-50 lbs.; heavy (yellow color) with resistance 7 (R7) 0-70 lbs. All subjects completed three study visits, and a total of four measurements were taken at baseline, immediately following the first session, at two weeks, and at 4 weeks.
  Arms: Sport cords

SUMMARY:
ProtonicsTM Knee brace has been suggested as an intervention for patients with patellofemoral pain syndrome (PFPS). However, the effectiveness of this knee brace compared to traditional conservative methods knee rehabilitation is lacking. The objective of this randomized controlled trial was to compare the effect of ProtonicsTM knee brace vs. sports cord on knee pain and function in patients with PFPS.

DETAILED DESCRIPTION:
The purpose of this graduate student research study was to compare the effect of ProtonicsTM knee brace vs. sports cord on knee pain and function in patients with PFPS.

Design: Randomized controlled trial.

Setting: Loma Linda University.

Participants: Subjects with patellofemoral pain will participate in the study.

Intervention: Subjects will be randomized to one of two treatment groups, the ProtonicsTM knee brace or the sport cord to complete a series of resistance exercises over the course of 4 weeks.

Main Outcome Measures: Both groups will be evaluated according to the following clinical outcomes: Anterior pelvic tilt (APT), hip internal/external rotation, and iliotibial band flexibility. The following functional outcomes were also assessed: Global Rating of Change (GROC) scale, the Kujala score, the Numeric Pain Rating Scale, and the lateral step-down test.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be males and females who have Patellofemoral pain symptoms for more than 1 month, have pain level ≥ 3 on a Numeric Pain Rating Scale, and pain during at least 2 activities, such as squatting, ascending/descending stairs, and/or running.

Exclusion Criteria:

* Subjects will be excluded if they have previous traumatic injuries to the knee joint/lower limbs, sign, and symptoms of meniscus tear or ligamentous-related pathology, neurological disorders and being on pain medication."

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Everett Lohman, Dsc, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arroll B, Ellis-Pegler E, Edwards A, Sutcliffe G. Patellofemoral pain syndrome. A critical review of the clinical trials on nonoperative therapy. Am J Sports Med. 1997 Mar-Apr;25(2):207-12. doi: 10.1177/036354659702500212. PMID 9079175
- [Result] Bockrath K, Wooden C, Worrell T, Ingersoll CD, Farr J. Effects of patella taping on patella position and perceived pain. Med Sci Sports Exerc. 1993 Sep;25(9):989-92. PMID 8231783
- [Result] Callaghan MJ, Selfe J. Patellar taping for patellofemoral pain syndrome in adults. Cochrane Database Syst Rev. 2012 Apr 18;2012(4):CD006717. doi: 10.1002/14651858.CD006717.pub2. PMID 22513943
- [Result] Azevedo DC, Santos H, Carneiro RL, Andrade GT. Reliability of sagittal pelvic position assessments in standing, sitting and during hip flexion using palpation meter. J Bodyw Mov Ther. 2014 Apr;18(2):210-4. doi: 10.1016/j.jbmt.2013.05.017. Epub 2013 Jun 17. PMID 24725788
- [Result] Denton J, Willson JD, Ballantyne BT, Davis IS. The addition of the Protonics brace system to a rehabilitation protocol to address patellofemoral joint syndrome. J Orthop Sports Phys Ther. 2005 Apr;35(4):210-9. doi: 10.2519/jospt.2005.35.4.210. PMID 15901122
- [Result] Earl JE, Piazza SJ, Hertel J. The Protonics Knee Brace Unloads the Quadriceps Muscles in Healthy Subjects. J Athl Train. 2004 Mar;39(1):44-49. PMID 15085211
- [Result] Gajdosik RL, Sandler MM, Marr HL. Influence of knee positions and gender on the Ober test for length of the iliotibial band. Clin Biomech (Bristol). 2003 Jan;18(1):77-9. doi: 10.1016/s0268-0033(02)00168-7. PMID 12527250

RESULTS

PARTICIPANT FLOW:
Groups:
- Protonics Knee Brace: All subjects were fitted with a regular-sized Protonics knee brace with resistive settings to resist knee flexion.
  Protonics Knee brace: Protonics Therapy Program is separated into three phases for a period of 4 weeks. In each phase the patients will learn how to perform the Protonics neuromuscular repositioning technique, Protonics gait and open-chain exercise. All subjects will be asked to perform the exercise 3 times a week, 3 sets a day; every set is 10-15 repetitions for 4 weeks In phase one, the subjects will perform Protonics Neuromuscular repositioning Techniques, Protonics gait through walking for up to 5 minutes or as tolerated, and preform warming up exercise.
  In phase two, the subjects will perform Protonics Neuromuscular repositioning Techniques, Protonics gait through walking for up to 8 minutes or as tolerated, and preform three specific exercises in prone, supine and sitting position.
  In phase three, the subjects will perform Protonics exercises.
- Sport Cords: Resistive sports cord to resist knee flexion.
  Sports Cords: Sports Cord Therapy Program is separated into three phases for a period of 4 weeks. In each phase the patients will learn how to perform the sports cord gait and open-chain exercise. All subjects will be asked to perform the exercise 3 times a week, 3 sets a day; every set is 10-15 repetitions for 4 weeks.
  In phase one, the subjects will perform the sports cord gait through walking for up to 5 minutes or as tolerated, and preform warming up exercise.
  In phase two, the subjects will perform the sports cord gait through walking for up to 8 minutes or as tolerated, and preform three specific exercises in prone, supine and sitting position.
  In phase three, the subjects will perform the sports cord gait through walking for up to 10 minutes or as tolerated, and preform one specific exercise in standing position.
Period: Overall Study
Arm/Group | Protonics Knee Brace | Sport Cords
Started | 22 | 21
Completed | 21 | 20
Not Completed | 1 | 1
Not completed — drop out | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Protonics Knee Brace: Subjects were fitted with a regular-sized Protonics knee brace with resistive settings to resist knee flexion.
  Protonics Knee brace: Program was separated into three phases for a period of 4 weeks. Each phase the patients learned how to perform the Protonics neuromuscular repositioning technique, Protonics gait and open-chain exercise. Subjects asked to perform the exercise 3 times a week, 3 sets a day; every set is 10-15 repetitions for 4 weeks.
  Phase one, Subjects performed Protonics Neuromuscular repositioning Techniques, walking for up to 5 minutes or as tolerated, and preform warming up exercise.
  Phase two, subjects performed Protonics Neuromuscular repositioning Techniques, walking for up to 8 minutes or as tolerated, and preform three specific exercises in prone, supine and sitting position.
  Phase three, the subjects performed Protonics Neuromuscular repositioning Techniques, walking for up to 10 minutes or as tolerated, and preformed exercise in standing position.
- Total: Total of all reporting groups
Arm/Group | Protonics Knee Brace | Sport Cords | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 20 | 41
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (5.6) | 26.7 (3) | 28.81 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 9 | 12 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Anterior Pelvic Tilt
Description: Anterior Pelvic Tilt: tilting of the pelvic will be measured with CHEK inclinometer. Tilting will be measured while subjects are in a standing position. The examiner will determine the two measure line marks, anterior superior iliac spine (ASIS) and posterior superior iliac spine (PSIS) to find the oblique angle of the pelvic.
  Normative values from other study that we will be using to compare anterior pelvic tilt: Male = 9° and Female = 12° (from Nguyen study in 2007).
  The CHEK inclinometer caliper has two arms; one arm will be placed on ASIS (front of pelvis) while the other on the PSIS (back of pelvis). The angle of the caliper will be determined to record the degree of anterior pelvic tilt.
  Baseline measurement to Post-intervention measurement = Four (4) weeks.
Time Frame: Baseline to Post intervention
Measure: Mean (Standard Deviation); unit: degree
Groups:
- Protonics Knee Brace: All subjects were fitted with a regular-sized Protonics knee brace with resistive settings to resist knee flexion.
  Protonics Knee brace: Protonics Therapy Program is separated into three phases for a period of 4 weeks. In each phase the patients will learn how to perform the Protonics neuromuscular repositioning technique, Protonics gait and open-chain exercise. All subjects will be asked to perform the exercise 3 times a week, 3 sets a day; every set is 10-15 repetitions for 4 weeks In phase one, the subjects will perform Protonics Neuromuscular repositioning Techniques, Protonics gait through walking for up to 5 minutes or as tolerated, and preform warming up exercise.
  In phase two, the subjects will perform Protonics Neuromuscular repositioning Techniques, Protonics gait through walking for up to 8 minutes or as tolerated, and preform three specific exercises in prone, supine and sitting position.
  In phase three, the subjects will perform Protonics Neuromuscular repositioni
Arm/Group | Protonics Knee Brace | Sport Cords
Number analyzed (Participants) | 21 | 20
degree | 5 (2.8) | 3.2 (2.8)
Statistical Analysis 1: Comparison: Protonics Knee Brace vs Sport Cords; Data analysis was performed using SPSS Statistics Software version 24.0. We compared mean age (years), Body Mass Index (kg/m2) (BMI), pain duration, and the outcome measures at baseline in both groups at baseline using independent t-test when the distribution of the variable was approximately normal and Mann-Whitney test when the distribution was not normal. The distribution of qualitative variables (gender, affected leg) by group type was examined using Chi Square test; Test type: Superiority; Wilcoxon (Mann-Whitney) — a priori threshold for statistical significance is <0.05; a priori threshold for statistical significance is <0.05

2. Primary Outcome: Anterior Pelvic Tilt
Description: Anterior Pelvic Tilt: tilting of the pelvic will be measured with CHEK inclinometer. Tilting will be measured while subjects are in a standing position. The examiner will determine the two measure line marks, anterior superior iliac spine (ASIS) and posterior superior iliac spine (PSIS) to find the oblique angle of the pelvic. Approximate normally anterior pelvic tilt for male is 9° and for female is about 12° (Nguyen, 2007). The caliper has two arms; one arm will be placed on ASIP while the other on the PSIS. The angle of the caliper will be determined to record the degree of anterior pelvic tilt.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Protonics Knee Brace | Sport Cords
Number analyzed (Participants) | 21 | 20
degree | 3.1 (2) | 2.5 (2)

3. Primary Outcome: Anterior Pelvic Tilt
Description: as for outcome 2
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Protonics Knee Brace | Sport Cords
Number analyzed (Participants) | 21 | 20
degree | 2 (1.6) | 1.9 (1.6)

4. Primary Outcome: Numeric Pain Rating Scale (NPRS)
Description: The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Protonics Knee Brace | Sport Cords
Number analyzed (Participants) | 21 | 20
cm | 4.5 (1.2) | 3.8 (1.9)

5. Primary Outcome: Numeric Pain Rating Scale (NPRS)
Description: Used to assess pain level throughout the intervention. Scale: 0-10. Scoring: 0 (no pain) to 10 (worst, imaginable pain).
Time Frame: Immediately following 1st session
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Protonics Knee Brace | Sport Cords
Number analyzed (Participants) | 21 | 20
cm | 3 (1.9) | 3.2 (1.9)

6. Primary Outcome: Numeric Pain Rating Scale (NPRS)
Description: as for outcome 4
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Protonics Knee Brace | Sport Cords
Number analyzed (Participants) | 21 | 20
cm | 1.9 (1.7) | 2.5 (1.7)

7. Primary Outcome: Numeric Pain Rating Scale (NPRS)
Description: Used to assess pain level throughout the intervention. Scale: 0-10. Scoring: 0 (no pain) to 10 (worst, imaginable pain).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Protonics Knee Brace | Sport Cords
Number analyzed (Participants) | 21 | 20
cm | 1.1 (1.7) | 2 (1.7)

8. Primary Outcome: Global Rating of Change (GROC)
Description: GROC scales offer a flexible, quick, and simple method of charting self-assessed clinical progress in research and clinical settings. 15-Point: Scale -7 to 0 to +7. A score of 0 = No change, +1 to +3 = small positive change, +4 to +5 = Moderate positive change, +6 to +7 = Large positive change. All negative scores (minus numbers) represent a poor outcome (-7 being the worst possible outcome).
Time Frame: Immediately following 1st session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Protonics Knee Brace | Sport Cords
Number analyzed (Participants) | 21 | 20
units on a scale | 1 (2.1) | 0 (2.1)
Statistical Analysis 1: Comparison: Protonics Knee Brace vs Sport Cords; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

9. Primary Outcome: Global Rating of Change (GROC)
Description: GRC scales offer a flexible, quick, and simple method of charting self-assessed clinical progress in research and clinical settings. It ranges from -7 to 7, in which item -7 represent very great deal worse, 0 represent no change in progress, and 7 exemplify a very great better.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Protonics Knee Brace | Sport Cords
Number analyzed (Participants) | 21 | 20
units on a scale | 3 (2.2) | 1.3 (2.2)

10. Primary Outcome: Global Rating of Change (GROC)
Description: as for outcome 9
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Protonics Knee Brace | Sport Cords
Number analyzed (Participants) | 21 | 20
units on a scale | 4.6 (2.3) | 3 (2.3)

11. Primary Outcome: Kujala Score
Description: A self-report questionnaire, which is used to evaluate subjective symptoms and functional limitations in subjects with PFPS with a score range between of 0 - 100 based on pain associated with variety of functional activities such as prolonged sitting, squatting, running, and jumping. A score close to 100 indicates a higher functional performance. A score close to 0 represents a low level of function. Kujala scale has shown acceptable test-retest reliability (rho = 0.86) (Paxon et al, 2003). Kujala scale scores will be documented at the beginning and end of the intervention program.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Protonics Knee Brace | Sport Cords
Number analyzed (Participants) | 21 | 20
points | 74.8 (12.1) | 79.3 (12.1)

12. Primary Outcome: Kujala Score
Description: A self-report questionnaire, which is used to evaluate subjective symptoms and functional limitations in subjects with PFPS with a score range between of 0 - 100 based on pain associated with variety of functional activities such as prolonged sitting, squatting, running, and jumping. A score close to 100 indicates a higher functional performance. Kujala scale has shown acceptable test-retest reliability (rho = 0.86) (Paxon et al, 2003). Kujala scale scores will be documented at the beginning and end of the intervention program.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Protonics Knee Brace | Sport Cords
Number analyzed (Participants) | 21 | 20
points | 87.5 (15.1) | 87.5 (15.1)

13. Primary Outcome: Lateral Step-Down Test
Description: Lateral step test: is a quick and simple practical clinical measure of functional. Subjects with PFPS will be asked to step up and down on a 15-cm step for 15 seconds each with a cadence of 2 steps per second. The total number of step-ups during this time will be recorded. Subjects will be asked to report a verbal pain score during the step-up test at each test session. This test will be performed every two weeks to document any improvement in the functional performance. The test has shown to be reliable and valid, with test-retest reliability of (ICC = 0.90) (Ross et al, 1997).
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Protonics Knee Brace | Sport Cords
Number analyzed (Participants) | 21 | 20
steps | 7 (2.7) | 9.1 (2.7)

14. Primary Outcome: Lateral Step-Down Test
Description: as for outcome 13
Time Frame: Immediately following 1st session
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Protonics Knee Brace | Sport Cords
Number analyzed (Participants) | 21 | 20
steps | 9.6 (3.3) | 11.8 (3.3)

15. Primary Outcome: Lateral Step-Down Test
Description: Lateral step test: is a quick and simple practical clinical measure of functional. Subjects with PFPS will be asked to step up and down on a 15-cm step for 15 seconds each with a cadence of 2 steps per second. The total number of step-ups during this time will be recorded. This test will be performed every two weeks to document any improvement in the functional performance. The test has shown to be reliable and valid, with test-retest reliability of (ICC = 0.90) (Ross et al, 1997).
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Protonics Knee Brace | Sport Cords
Number analyzed (Participants) | 21 | 20
steps | 13.3 (3.2) | 14.7 (3.2)

16. Primary Outcome: Lateral Step-Down Test
Description: as for outcome 15
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Protonics Knee Brace | Sport Cords
Number analyzed (Participants) | 21 | 20
steps | 16.3 (3.3) | 16.8 (3.3)

17. Secondary Outcome: Iliotibial Band Flexibility
Description: To assess the flexibility of iliotibial band
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Protonics Knee Brace | Sport Cords
Number analyzed (Participants) | 21 | 20
degree | 3.5 (2.7) | 3.2 (2.7)

18. Secondary Outcome: Iliotibial Band Flexibility
Description: To assess the flexibility of iliotibial band
Time Frame: Immediately following 1st session
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Protonics Knee Brace | Sport Cords
Number analyzed (Participants) | 21 | 20
degree | 2.1 (2.3) | 2.5 (2.3)

19. Secondary Outcome: Iliotibial Band Flexibility
Description: To assess the flexibility of iliotibial band
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Protonics Knee Brace | Sport Cords
Number analyzed (Participants) | 21 | 20
degree | 2.8 (1.9) | 1.8 (1.9)

20. Secondary Outcome: Iliotibial Band Flexibility
Description: To assess the flexibility of iliotibial band
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Protonics Knee Brace | Sport Cords
Number analyzed (Participants) | 21 | 20
degree | 0.4 (2.2) | 12 (2.2)

21. Secondary Outcome: Hip Internal Rotation ROM
Description: To measure the internal rotation of hip in sitting natural position with hip and knee on 90 degree flexion
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Protonics Knee Brace | Sport Cords
Number analyzed (Participants) | 21 | 20
degree | 25.9 (7) | 28.8 (7)

22. Secondary Outcome: Hip Internal Rotation ROM
Description: To measure the internal rotation of hip in sitting natural position with hip and knee on 90 degree flexion
Time Frame: Immediately following 1st session
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Protonics Knee Brace | Sport Cords
Number analyzed (Participants) | 21 | 20
degree | 25.5 (5.5) | 29.3 (5.5)

23. Secondary Outcome: Hip Internal Rotation ROM
Description: To measure the internal rotation of hip in sitting natural position with hip and knee on 90 degree flexion
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Protonics Knee Brace | Sport Cords
Number analyzed (Participants) | 21 | 20
degree | 29.2 (5) | 31.6 (5)

24. Secondary Outcome: Hip Internal Rotation ROM
Description: To measure the internal rotation of hip in sitting natural position with hip and knee on 90 degree flexion
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Protonics Knee Brace | Sport Cords
Number analyzed (Participants) | 21 | 20
degree | 29.4 (5.8) | 32.6 (5.8)

25. Secondary Outcome: Hip External Rotation ROM
Description: To measure the External rotation of hip in sitting natural position with hip and knee on 90 degree flexion
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Protonics Knee Brace | Sport Cords
Number analyzed (Participants) | 21 | 20
degree | 31.3 (4.9) | 31.3 (4.9)

26. Secondary Outcome: Hip External Rotation ROM
Description: To measure the External rotation of hip in sitting natural position with hip and knee on 90 degree flexion
Time Frame: Immediately following 1st session
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Protonics Knee Brace | Sport Cords
Number analyzed (Participants) | 21 | 20
degree | 32.2 (5) | 32.5 (5)

27. Secondary Outcome: Hip External Rotation ROM
Description: To measure the external rotation of hip in sitting natural position with hip and knee on 90 degree flexion
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Protonics Knee Brace | Sport Cords
Number analyzed (Participants) | 21 | 20
degree | 32.3 (5.2) | 32.3 (5.2)

28. Secondary Outcome: Hip External Rotation ROM
Description: To measure the external rotation of hip in sitting natural position with hip and knee on 90 degree flexion
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Protonics Knee Brace | Sport Cords
Number analyzed (Participants) | 21 | 20
degree | 33.9 (5.7) | 33.9 (5.7)

ADVERSE EVENTS:
Time Frame: The study has concluded. During the entire 4-week experiment (baseline to conclusion), no adverse event (AEs) occurred to any of the subjects. Subjects participated in one of two exercise programs over a 4 week period from baseline testing to the conclusion of the study. In each group, exercises were to be performed 3 times per week. This represents a total 12 exercise sessions (3 x 4 WEEKS ). Each session included 3 sets of 10-15 repetitions for each exercise as outlined.
Groups:
- Protonics Knee Brace: All subjects were fitted with a regular-sized Protonics knee brace with resistive settings to resist knee flexion.
  Protonics Knee brace: Protonics Therapy Program is separated into three phases for a period of 4 weeks. All subjects will be asked to perform the exercise 3 times a week, 3 sets a day; every set is 10-15 repetitions for 4 weeks. Subjects will be monitored for any and all adverse events including excessive Delayed Onset Muscle Soreness throughout the study during the three (3) phases of the .
  Protonics Neuromuscular repositioning Technique training,
- Sport Cords: Resistive sports cord to resist knee flexion.
  Sports Cords: Sports Cord Therapy Program is separated into three phases for a period of 4 weeks. In each phase the patients will learn how to perform the sports cord gait and open-chain exercise. All subjects will be asked to perform the exercise 3 times a week, 3 sets a day; every set is 10-15 repetitions for 4 weeks.Subjects will be monitored for any and all adverse events including excessive Delayed Onset Muscle Soreness throughout the study during the three (3) phases of the Sport Cord training,
Arm/Group | Protonics Knee Brace | Sport Cords
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/21 | 0/20

LIMITATIONS AND CAVEATS:
The intervention protocol was only four weeks, which is a short time period, and it is possible that with a longer study duration, differences between the intervention groups may have become more evident.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-11): https://cdn.clinicaltrials.gov/large-docs/59/NCT03042559/Prot_SAP_000.pdf